CLINICAL TRIAL: NCT07151053
Title: Validity and Reliability of the Duruöz Hand Index in Obstetric Brachial Plexus Palsy
Brief Title: Duruöz Hand Index in Obstetric Brachial Plexus Palsy
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Bilal Kulaksiz, Physical medicine and rehabilitation specialist, Istanbul University - Cerrahpasa
Other Study IDs: 83045809-604.01.02-
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Obstetric Brachial Plexus Injury
Keywords: Brachial plexus; Duruöz Hand Index

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Grup 1: The study included twenty-one children aged 6 to 18 years, all diagnosed with OBPP, who were followed up at the Physical Medicine and Rehabilitation outpatient clinic of a tertiary university hospital in Turkey. The exclusion criteria were a history of trauma or surgery affecting the function of the affected extremity (other than OBPP), the presence of systemic diseases that could impair hand function (such as polyneuropathy), and cognitive impairments that could affect comprehension.

SUMMARY:
Obstetric brachial plexus palsy (OBPP) arises from perinatal injury to the brachial plexus, resulting in varying degrees of motor and sensory impairment in the upper extremity. While existing assessment instruments primarily target unilateral limb function, they frequently overlook bimanual capabilities, which are essential for functional independence. This study aims to investigate the utility of the Duruöz Hand Index (DHI) as a reliable, valid, and practical instrument for evaluating functional limitations in individuals with OBPP. A cohort of 21 pediatric patients (aged 6-18 years) with OBPP was recruited from a tertiary university hospital in Turkey. Functional assessment included grip and pinch strength, range of motion, and upper extremity performance, measured using the Modified Mallet Classification, Brachial Plexus Outcome Measure (BPOM), Pediatric Outcomes Data Collection Instrument (PODCI), and DHI

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 18 years
* All diagnosed with OBPP who were followed up at the Physical Medicine and Rehabilitation outpatient clinic of a tertiary university hospital in Turkey.

Exclusion Criteria:

* A history of trauma or surgery affecting the function of the affected extremity (other than OBPP)
* The presence of systemic diseases that could impair hand function (such as polyneuropathy)
* Cognitive impairments that could affect comprehension.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study cohort consisted of patients who were under regular follow-up at our tertiary care hospital and met the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Validity and reliability | At baseline
  The primary outcome measure was the Duruöz Hand Index (DHI), which was investigated to determine whether it can adequately capture impairments in bimanual function during daily activities and provide a comprehensive assessment of functional disability in patients with OBPP. To evaluate the validity of the DHI, its correlations with established outcome measures-including the Modified Mallet Classification, Brachial Plexus Outcome Measure (BPOM), Pediatric Outcomes Data Collection Instrument (PODCI), as well as grip and pinch strength and range of motion-were examined. Reliability was assessed through internal consistency using Cronbach's alpha.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğçe Özekli Mısırlıoğlu, Prof., PM&R, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) collected during this study will be shared in an anonymized format. All identifying information will be removed to ensure participant confidentiality, and only de-identified datasets underlying the study results will be made available to qualified researchers upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: De-identified individual participant data (IPD) and supporting documents will be available starting from the date of publication of the main study results and will remain accessible for 5 years.
Access Criteria: IPD and supporting information will be accessible to qualified researchers for academic or scientific purposes. Access requests can be submitted via email to the corresponding author, and data will be shared after approval and signing of a data use agreement to ensure confidentiality and ethical use.

REFERENCES:
- [Background] Misirlioglu TO, Unalan H, Karamehmetoglu SS. Validation of Duruoz Hand Index in patients with tetraplegia. J Hand Ther. 2016 Jul-Sep;29(3):269-74. doi: 10.1016/j.jht.2015.10.001. Epub 2015 Oct 22. PMID 26541579
- [Background] Duruoz MT, Poiraudeau S, Fermanian J, Menkes CJ, Amor B, Dougados M, Revel M. Development and validation of a rheumatoid hand functional disability scale that assesses functional handicap. J Rheumatol. 1996 Jul;23(7):1167-72. PMID 8823687
- [Background] O'Berry P, Brown M, Phillips L, Evans SH. Obstetrical Brachial Plexus Palsy. Curr Probl Pediatr Adolesc Health Care. 2017 Jul;47(7):151-155. doi: 10.1016/j.cppeds.2017.06.003. Epub 2017 Jul 12. PMID 28709767